CLINICAL TRIAL: NCT07154641
Title: Comparison Between Latissimus Dorsi Tendon Transfer and Superior Capsular Reconstruction in Massive Rotator Cuff Tears: A Randomised Controlled Trial.
Brief Title: Latissimus Dorsi Tendon Transfer vs. Superior Capsular Reconstruction in Massive Rotator Cuff Tears
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konstantopoulio-Patission General Hospital of Nea Ionia (Other)
Responsible Party: Principal Investigator, Dimitrios V Papadopoulos, Assistant Professor of Orthopaedics, Konstantopoulio-Patission General Hospital of Nea Ionia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102/13-3-25
Record Dates: First submitted 2025-07-06; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Massive Rotator Cuff Tears
Keywords: Massive rotator cuff tears; Latissimus dorsi tendon transfer; Superior capsular reconstruction; rotator cuff tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latissimus dorsi tendon transfer group (Active Comparator): 22 patients are expected to undergo latissimus dorsi tendon transfer for the treatment of massive rotator cuff tears
  Interventions: Procedure: Latissimus dorsi tendon transfer
- Superior capsular reconstruction group (Active Comparator): 22 patients are expected to undergo superior capsular reconstruction for the treatment of massive rotator cuff tears.
  Interventions: Procedure: Superior capsular reconstruction

INTERVENTIONS:
Procedure: Latissimus dorsi tendon transfer — Latissimus dorsi tendon transfer is a surgical procedure that aims to restore active range of motion and stability of the shoulder in patients with massive rotator cuff tears. The tendon of the latissimus dorsi muscle is dettached from its insertion in the midbicipital groove of the humerus and reattached to the greater tubetosity. Therefore, the muscle acts as an external rotator, while the forces created pull the humeral head down and stabilize it in the glenoid.
  Arms: Latissimus dorsi tendon transfer group
Procedure: Superior capsular reconstruction — Superior capsular reconstruction is a surgical procedure that aims to restore shoulder stability in patients with massive rotator cuff tears. The superior capsule of the shoulder joint is attached to the greater tuberosity and is therefore often torn in cases of supraspinatus or infraspinatus tears. A fascia lata autograft is used to reconstruct the torn capsule, between the greater tuberosity and the glenoid. Thus, superior migration of the humeral head is prevented, and pain and functionality are improved.
  Arms: Superior capsular reconstruction group

SUMMARY:
The goal of this clinical trial is to compare the results of two surgical operations for the treatment of massive rotator cuff tears: latissimus dorsi tendon transfer (LDT) and superior capsular reconstruction (SCR).

The main question it wants to answer is which of the two operations provides better functional results, as measured by two patient-reported questionaires: the American Shoulder and Elbow Surgeons (ASES) score and the Constant-Murley score.

The patients will be randomly assigned to one of two groups according to the surgery they will undergo (LDT or SCR). They will be examined clinically and asked to fill the questionaires before the surgery, at 6 weeks and at 3, 6, 12 and 24 months after surgery.

DETAILED DESCRIPTION:
The participants will be included in the research protocol by Mai 2025. The sample size is determined through a power analysis based on the postoperative Constant scores of a similar trial after 31 months of follow-up (see References). Τhe mean difference between preoperative and postoperative Constant scores was used to calculate sample size with a power of 80% and a=0.05. A two-tailed test was used for two independent mean values with effect size d=0.8841. According to the power analysis, 22 patients are required for each cohort (44 patients in total) to achieve a statistically significant difference between mean preoperative and postoperative Constant scores. The critical t value was 2.018 for 42 degrees of freedom. The authors used the Shapiro-Wilk test to confirm the normal distribution of the data. The power analysis was conducted using the G*power 3.1 software. Enrolled patients will be randomized into two treatment cohorts by a member of the research team who will be blinded to the preoperative patient data, with randomization software. 22 patients will undergo latissimus dorsi tendon transfer (LDT) and 22 patients will undergo superior capsular reconstruction (SCR).

Primary outcomes include the Constant score, the American Shoulder and Elbow Surgeons (ASES) score, and the Visual Analog Scale (VAS) for pain assessment. Secondary outcomes include the progression to osteoarthritis, the measurement of the acromiohumeral distance (AHD) and the treatment of pseudoparalysis.

The patients will be physically examined before surgery, at 6 weeks and at 3 months, 6 months, 12 months and 24 months after surgery. During follow-ups in 3, 6, 12 and 24 months postoperatively, patients will be physically examined by a member of the research team who will be blinded to the type of surgery.

To assess active range of motion (ROM) in forward flexion, abduction, internal and external rotation, a typical goniometer will be used. Patients should be upright with the scapula stabilised in the vertical plane. Additionally, muscle strength will be assessed using a handheld dynamometer. Patients will fill in the Constant, ASES and VAS questionnaires in each follow-up. Moreover, in 2, 12 and 24 months after surgery anterior-posterior radiographs will be performed. Radiographs will be assessed for the progression of rotator cuff arthropathy (based on the Hamada classification) and the AHD will be measured by a radiologist who will be blinded to the type of surgery.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (over 18 years old). Massive rotator cuff tear diagnosis based on shoulder MRI. -

Exclusion Criteria:

Advanced glenohumeral arthritis (Hamada ≥3). Deltoid dysfunction. Irrepearable subscapularis tear. Infection. Prior shoulder surgery. Shoulder stiffness.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Constant-Murley score | Before surgery, at 6 weeks and at 3, 6, 12, and 24 months after surgery, per participant.
  Functionality will be measured based on the Constant-Murley score. This questionaire includes 4 sections, regarding pain, activities of daily living (ADL), range of motion (ROM) and muscle strength. The questions regarding pain and ADL are filled by the patients, whereas the assessment of ROM and muscle strength require physical examination by a member of the research team. For the assessment of strength a handheld dynamometer will be used. The minimum score is 0 and the maximum 100.
American Shoulder and Elbow Surgeons (ASES) score | Before surgery, at 6 weeks and at 3, 6, 12, and 24 months after surgery, per participant.
  American Shoulder and Elbow Surgeons (ASES) score, measures functionality of the shoulder. It includes 17 multiple-choice questions which are filled by the patients and is divided in two sections: one section about pain assessment and one about activities of daily living (ADL). The minimum score is 0 and the maximum 100.
Visual Analog Scale (VAS) for pain | Before surgery, at 6 weeks and at 3, 6, 12, and 24 months after surgery, per participant.
  The Visual Analog Scale for pain is a scale from 0 to 10, that measures the intensity of pain and is a patient-reported score. 0 means "no pain at all" and 10 "pain as bad as it can be". The scale is included in the Pain Questionaire of the American Shoulder and Elbow Surgeons (ASES) score.
Active Range of Motion (ROM) | Before surgery, at 6 weeks and at 3, 6, 12, and 24 months after surgery, per participant.
  The active Range of Motion (ROM) will be measured before and after surgery and compared between the two arms. The participants will be examined clinically by an investigator who will be blinded to the type of surgery. The active ROM in forward flexion, abduction, internal and external roation of the shoulder will be examined. For this purpose, a typical goniometer will be used. During the examination the patients should be standing and the scapula should be stabilised in the vertical plane.
Muscle strength | Before surgery, at 6 weeks and at 3, 6, 12, and 24 months after surgery, per participant.
  Muscle strength will be measured using a hand dynamometer. This is included in the last section of the Constant-Murley score. Minimum score is 0 and maximum is 25. The score is calculated as 1 point per pound or 2.2 points per kilogram. The patient should hold the weight with the arm in 90° of abduction and the elbow extended for at least 3 seconds. Three consecutive measurements are performed with at least 1 minute break in between. The measurement with the best score defines the overall score. If the patients are unable to abduct the arm 90° or if they are experiencing pain, the score is 0.

SECONDARY OUTCOMES:
Treatment of Pseudoparalysis | Before surgery, at 6 weeks and at 3, 6, 12, and 24 months after surgery, per participant.
  Pseudoparalysis is defined as inability of forward flexion at 90°, with absence of neurological deficit, and maintained passive range of motion (ROM). Patients will be examined clinically for the progression or treatment of pseudoparalysis and the results will be compared between the two arms.
Progression of Rotator Cuff Arthropathy | Before surgery, at 6 weeks and at 3, 6, 12, and 24 months after surgery, per participant.
  The progression of rotator cuff arthropathy will be assessed. by a radiologist who will be blinded to the type of treatment. Radiographs will be taken at 2, 12 and 24 months after surgery and the progression of osteoarthritis will be examined based on the Hamada classification (grade I to V). The acromiohumeral distance will also be measured in each radiograph. The results will be compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios V Papadopoulos, MD, PhD, Principal Investigator — Second Department of Orthopaedics, Medical School, National and Kapodistrian University of Athens, Athens, Greece
Locations (1):
- Konstantopouleio-Patision General Hospital of Nea Ionia, Athens, Attica, Greece

REFERENCES:
- [Background] Ozturk BY, Ak S, Gultekin O, Baykus A, Kulduk A. Prospective, randomized evaluation of latissimus dorsi transfer and superior capsular reconstruction in massive, irreparable rotator cuff tears. J Shoulder Elbow Surg. 2021 Jul;30(7):1561-1571. doi: 10.1016/j.jse.2021.01.036. Epub 2021 Mar 4. PMID 33675971